CLINICAL TRIAL: NCT05057078
Title: The Effect of Mindfulness-Based Stress Reduction Program on Spiritual Well-being in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: The Effect of Mindfulness Program on Spiritual Well-BeingBreast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice ÖNER CENGİZ, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OnerCengiz
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Nursing Caries
Keywords: Breast cancer; Spirituality; Nursing Care; Mindfulness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A mindfulness-based stress reduction program will be done once a week for eight weeks
  Interventions: Behavioral: mindfulness-based stress reduction program
- Control group (No Intervention): During study process, no application will be made to the control group.

INTERVENTIONS:
Behavioral: mindfulness-based stress reduction program — groups of 10 people will be formed among the patients included in the mindfulness program group. A mindfulness-based stress reduction program will be done once a week for eight weeks and will take approximately 60-120 minutes. A plan will be made with the patients for the day and time of the session. During this process, no application will be made to the control group. Meetings will be held as an online session via Zoom Video Communications.
  Arms: Intervention group

SUMMARY:
Breast cancer ranks first among the cancers seen in women in the World. Due to breast cancer, patients experience spiritual distress. The aim of this study is to determine the effect of mindfulness-based stress reduction program applied to patients with breast cancer on spiritual well-being.

DETAILED DESCRIPTION:
Breast cancer ranks first among the cancers seen in women in the world and in Turkey . Physical and psychological symptoms may occur in breast cancer depending on the disease or the treatment applied. These symptoms cause patients to be perceived as a life-threatening disease and decrease their quality of life. This situation can create a crisis situation by deeply affecting the physical, psychosocial, behavioral and spiritual aspects of patients. In such a case, the patient can start using spiritual coping methods by turning to spirituality while facing a painful illness. Patients diagnosed with breast cancer have difficulty in finding the meaning and purpose of life, question their previous beliefs about life, and their concerns about spirituality, both existential and religious, increase. Spiritual dimensions, which are an important component of the patient's quality of life, are an integral part of patient care. Spirituality is used as a means of coping with cancer by providing inner strength, peace, comfort and integrity and can play an important role in healing and having a good mood . Therefore, raising the spiritual well-being of women with breast cancer may have a positive effect on coping with the symptoms of the disease and treatment, thereby improving the quality of life. Studies have shown that patients with high spiritual well-being have a higher quality of life. In a systematic review, it was found that religion/spirituality is associated with pain and physical symptoms, and spiritual self-evaluation contributes to psychological well-being, regardless of religion. In recent studies with breast cancer patients, it has been determined that mindfulness therapy has a positive effect on the quality of life of patients in addition to spirituality. Mindfulness is a way of directing attention, coming from the eastern tradition of meditation. It can be defined as an individual's focusing his attention on what is happening now in a non-judgmental and accepting way. The concept of mindfulness has been used as a therapy method in Western psychotherapy approaches for almost three decades. The concept of mindfulness basically includes focusing on the moment and accepting emotions without judgment . It allows the person to stay in the moment by focusing their attention. Staying in the moment contributes to the well-being of mood by preventing the mind from focusing on the past or the future and preoccupying the mind with various emotions Kabat-Zinn (2005), one of the practitioners of conscious mindfulness therapy, stated that mindfulness is closely related to the spiritual traditions of Far Eastern countries. Efforts to use Mindful Awareness to improve psychological processes continue. No study has been found in the literature examining the effect of mindfulness therapy on the spiritual well-being of patients with breast cancer. However, there is a need for initiatives to increase spiritual well-being , which is known to have a significant impact on quality of life. Therefore, the aim of this study is to determine the effect of mindfulness-based stress reduction program applied to patients with breast cancer on spiritual well-being.

METHODS This study is a single center, pretest-posttest with control group controlled trial. Participants will recruite in department of radiation oncology and oncology outpatient clinic of a tertiary hospital in Malatya from October 15, 2021 to May 15, 2022. Permission for the study was obtained from the ethics committee (E-41901325-050.99-14950). Written, fully informed consent will obtain from all participants and all data will guaranteed to be confidential. Participants has the right to withdraw from the study at any time. This study will conduct in accordance with The Consolidated Standards of Reporting Trials (CONSORT) 2010 guidelines.

Participants and Sampling We used the G * Power (version 3.1.9.4) test to determine the sample size. In the analysis performed as a priori, we referenced the Park et al. (2020) article. We performed prior analyses based on t-tests (mean values: difference between two independent mean values (two groups)). According to this, we determined that a total of 66 patients, including 33 patients in each of the groups with 0.05 error level, 95% power and 0.90 effect size, should be included. Aynı çalışmada drop out oranı %7.8 bulunmuştur. Given the likelihood of withdrawals, we will assign 35 participants to each group, with a total of 70 participants.

Randomization and blinding The participants will assign randomly to the groups. The simple full randomization method will use for group assignments. To determine the order of application, the names of the study groups (mindfulness program group and control group) will write on a piece of paper 30 times by the researcher, and the groups will select randomly by drawing lots. It will not possible for the researcher collecting data to be blind.

Data collection In data collection, the Socio-demographic Characteristics Form prepared by the researchers in line with the literature to determine the sociodemographic characteristics of the patients and the FACIT-SP (Functional Evaluation of the Treatment of Chronic Diseases-Spiritual Well-being) scale will be used to determine the spiritual well-being of the patients.

Socio-demographic Characteristics Form: This form, which was prepared by the researchers in line with the literature, consists of 18 questions includes patients' age, gender, marital status, education, employment status, occupation, presence of social security, income level, number of children, time of diagnosis, time to start treatment, stage of the disease, the presence of support in this disease, experiences that negatively affect thepatient, and methods of coping with them.

FACIT-Sp-Version 4: Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Scala FACIT-Sp-Version 4; It is a combined version of FACIT-G consisting of 4 sub-dimensions, 27 items, for quality of life assessment and FACIT-Sp-12, consisting of 3 sub-dimensions and 12 items, for spiritual assessment. The scale consists of 4 subscales, namely Physical Status (7 items), Social Life and Family Status (7 items), Emotional Status (6 items) and Activity Status (7 items) and a total of 27 items (http://www.facit .org-website). The Turkish validity and reliability study of the scale was carried out by Aktürk.et al. (2017). Cronbach's alpha values were determined to be 0.87 for the FACIT-Sp: 0.78 for the meaning subscale, 0.81 for the peace subscale, and 0.93 for the faith subscale.

Implementation of the initiative Before starting the study, the Socio-demographic Characteristics Form and the FACIT-SP (Functional Evaluation of the Treatment of Chronic Diseases-Spiritual Well-being) scale will be applied to the patients included in the mindfulness program group and control group in order to collect the pre-test data. After the pre-test data are collected, groups of 10 people will be formed among the patients included in the mindfulness program group. A mindfulness-based stress reduction program will be done once a week for eight weeks and will take approximately 60-90 minutes. A plan will be made with the patients for the day and time of the session. During this process, no application will be made to the control group. Meetings will be held as an online session via Zoom Video Communications. Post-test data will be collected from all patients after eight sessions. Each of the patients participating in the eight-week mindfulness-based stress reduction program will be retested 2 months after the program ends.

Statistical analysis Research data will be evaluated with the SPSS 25 (Statistical Package for Social Science) package program. Kolmogorov-Smirnov distribution test will be used to examine the normal distribution and Cronbach's alpha will be used for internal consistency. In the evaluation of the data, number, percentage, mean, standard deviation and parametric (t-test, analysis of variance) or nonparametric (Mann-Whitney U, Kruskal-Wallis tests) tests will be used according to the normal distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* Speaking and understanding Turkish,
* 18 to 65 year olds,
* diagnosed at least 6 months ago,
* Stage I, II or III breast cancer,
* To be receiving outpatient treatment,
* No barriers to joining online sessions.

Exclusion Criteria:

* Having a diagnosed psychiatric illness or disorder,
* End stage breast cancer,
* Refusing to participate in the study,
* Not participating regularly in the applied psycho-education program,
* Making a psychiatric diagnosis after the research has started,
* Initiation of inpatient treatment in the hospital.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
spiritual well-being-first | immediately before the first session
  The spiritual well-being level of the patients will be evaluated with FACIT-Sp scale
spiritual well-being-last | immediately after the last session
  The spiritual well-being level of the patients will be evaluated with FACIT-Sp scale

SECONDARY OUTCOMES:
Quality of life-first | immediately before the first session
  The quality of life level of the patients will be evaluated with FACIT-Sp scale
Quality of life-last | immediately after the last session
  The quality of life level of the patients will be evaluated with FACIT-Sp scale

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Öner Cengiz, PhD., Study Director — Ankara University
Locations (2):
- Turkey (Türkiye) (2):
  - Hatice ÖNER CENGİZ, Altındağ, Ankara
  - İnönü university Turgut Ozal Medicine Central, Malatya

REFERENCES:
- [Derived] Oner Cengiz H, Bayir B, Sayar S, Demirtas M. Effect of mindfulness-based therapy on spiritual well-being in breast cancer patients: a randomized controlled study. Support Care Cancer. 2023 Jul 3;31(7):438. doi: 10.1007/s00520-023-07904-2. PMID 37395841